CLINICAL TRIAL: NCT01902277
Title: ICU Delirium: a One-week Snapshot of Burden Across the Eastern UK Region
Status: Completed | Type: Observational
Sponsor: Papworth Hospital NHS Foundation Trust (Other Government)
Collaborators: Norfolk, Suffolk, and Cambridgeshire Critical Care Network (NSC CCN) (Unknown)
Responsible Party: Sponsor
Other Study IDs: P01535
Record Dates: First submitted 2013-07-15; First posted 2013-07-18 (Estimated); Last update posted 2013-07-18 (Estimated); Status verified 2013-07

CONDITIONS: Delirium
Keywords: Delirium; Intensive Care Unit; Critical illness
MeSH Terms: conditions — Delirium; Critical Illness

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Adult critically ill patients: All adult patients treated within study time frame on Intensive Care Units across Norfolk, Suffolk, and Cambridgshire, UK

SUMMARY:
ICU delirium negatively impacts on patient outcomes, as well as on resources and clinical workflow of the ICU. Effective healthcare resource planning requires reliable (i.e., multicentre) data that can inform on both of these.

The purpose of this study was to determine the impact of ICU delirium in terms of both patients and beds. The study was carried out prospectively, over a one-week period, at adult ICUs comprising the Norfolk, Suffolk, and Cambridgeshire Critical Care Network (NSC CCN).

DETAILED DESCRIPTION:
Previous delirium prevalence research has been carried out at single sites and yielded highly variable results (between 3-87%). Reliable multisite data can be obtained cost-effectively using a point-prevalence ("snapshot") approach.

Purpose: to obtain reliable data informing on prevalence of ICU delirium, in terms of both patients and beds, across the eastern UK region.

Design and Setting: this one-week observational prospective cohort study was carried out between June 25, 2012 (start of ICU day shift) to July 01, 2012 (end of night shift). Nine ICUs comprising the Norfolk, Suffolk, and Cambridgeshire Critical Care Network (NSC CCN) took part. Cambridgeshire 2 Research Ethics Committee approved the study (REC reference: 10/H0308/116) and waived the need for informed consent.

Patients and procedure: All adults treated over the study week at participating ICUs were considered eligible for inclusion. Delirium screening was carried out by patients' direct care clinicians using the Confusion Assessment Method for the ICU (CAM-ICU). All sites used this tool as part of their routine clinical practice and had delirium management guidelines in place at the time of the study. Patients who screened positive for delirium were treated according to local hospital practice.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients treated within study time frame on Intensive Care Units across Norfolk, Suffolk, and Cambridgshire, UK

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult critically ill patients across eastern UK region
Sampling Method: Probability Sample
Enrollment: 225 (Actual)
Dates: Start 2012-06; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Delirium prevalence | June 25, 2012 (start of ICU day shift) to July 1, 2012 (end of ICU night shift)
  Number of patients with at least one recorded delirium-positive result, over total number of patients recorded over study time frame. Delirium screening will be carried out using the CAM-ICU by local direct care clinicians in accordance with region-wide clinical delirium-screening guidelines.

SECONDARY OUTCOMES:
Proportion of patient-days with delirium | June 25, 2012 (start of ICU day shift) to July 1, 2012 (end of ICU night shift)
  Number of patient-days with at least one recorded delirium-positive result over total patient-days recorded.
Median delirium duration | June 25, 2012 (start of ICU day shift) to July 1, 2012 (end of ICU night shift)
  In delirium patients: median number of days recorded with delirium over study time frame.
Median days to transition to delirium | June 25, 2012 (start of ICU day shift) to July 1, 2012 (end of ICU night shift)
  In delirium patients admitted during study time frame: median number of days from ICU admission to first recorded delirium day.
Patient age, by delirium status | June 25 (start of ICU day shift) to July 1, 2012 (end of ICU night shift)
  In delirium patients versus patients with no recorded delirium-positive result over study time frame: median age.
Patient gender, by delirium status | June 25 (start of ICU day shift) to July 1, 2012 (end of ICU night shift)
  In delirium patients versus patients with no recorded delirium-positive result over study time frame: number of males over total patients in each group.
Admission type, by delirium status | June 25 (start of ICU day shift) to July 1, 2012 (end of ICU night shift)
  In delirium patients versus patients with no recorded delirium-positive result over study time frame: number of (1) urgent/emergency and (2) elective admissions, over total patients in each group.
Admission reason, by delirium status | June 25 (start of ICU day shift) to July 1, 2012 (end of ICU night shift)
  In delirium patients versus patients with no recorded delirium-positive result over study time frame: number of (1) medical and (2) surgical admissions, over total patients in each group.
Organ support, by delirium status | June 25 (start of ICU day shift) to July 1, 2012 (end of ICU night shift)
  In delirium patients versus patients with no recorded delirium-positive result over study time frame: number receiving advanced and basic respiratory, advanced and basic cardiovascular, and renal support since ICU admission to end of study time frame, over total patients in each group.
Mobilisation therapy, by delirium status | June 25 (start of ICU day shift) to July 1, 2012 (end of ICU night shift)
  In delirium patients versus patients with no recorded delirium-positive result over study time frame: number receiving mobilisation therapy over study time frame, over total patients in each group.
Median ICU days, by delirium status | June 25 (start of ICU day shift) to July 1, 2012 (end of ICU night shift)
  In delirium patients versus patients with no recorded delirium-positive result over study time frame: median number of patient-days in ICU per patient, since admission to end of study time frame.
Delirium screening compliance | June 25 (start of ICU day shift) to July 1, 2012 (end of ICU night shift)
  Number of patient-days CAM-ICU administered (1) once or more and (2) twice or more, over total number of patient-days recorded over study time frame.

CONTACTS AND LOCATIONS:
Overall Officials: Alain Vuylsteke, MD, Principal Investigator — Papworth Hospital NHS Foundation Trust
Locations (1):
- Papworth Hospital NHS Foundation Trust, Cambridge, Cambridgeshire, United Kingdom